CLINICAL TRIAL: NCT06460324
Title: Assessment of COVID-19 Vaccination Immune Response in Multiple Sclerosis Patients Treated With Ofatumumab in the United States: A Multicenter Medical Record Review Study
Brief Title: A Study to Assess COVID-19 Vaccination Immune Response in Multiple Sclerosis Patients Treated With Ofatumumab
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GUS27
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- COVID-19 Vaccination Cohort: Patients with multiple sclerosis (MS) who were receiving ofatumumab at the time of full COVID-19 vaccination and/or first booster vaccination.

SUMMARY:
This was a non-interventional, retrospective, observational cohort study involving the abstraction and review of pertinent data from medical records by participating physicians, who completed a customized electronic case report form hosted on the secure electronic data capture system.

ELIGIBILITY:
Inclusion criteria:

* Aged at least 18 years of age upon receipt of first COVID-19 vaccination.
* Fully vaccinated with any FDA-authorized COVID-19 vaccination.
* Diagnosed with MS.
* Receiving ofatumumab at the time of either (or both) of the following:

  1. Initial COVID-19 vaccination.
  2. Booster vaccination.
* Had a documented measurement of humoral response at least 2 weeks after completion of either (or both) of the following:

  1. Full COVID-19 vaccination course.
  2. Booster vaccine (among patients receiving ofatumumab at the time of the booster).

     Exclusion criteria:
* Received treatment with monoclonal antibodies to treat or prevent COVID-19 at any time between the first COVID-19 vaccination to within 6 months of the last COVID-19 vaccination (booster-inclusive).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Number of Ofatumumab-treated Patients with an Immune Response to FDA-authorized COVID-19 Vaccination by Vaccination Status | From 2 weeks up to 6 months post-vaccine
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
Number of Ofatumumab-treated Patients with an Immune Response to FDA-authorized COVID-19 Vaccination by Prior Disease Modifying Therapy (DMT) | From 2 weeks up to 6 months post-vaccine
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P.

SECONDARY OUTCOMES:
Mean Age at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Mean Age at Index Date by Prior Disease Modifying Therapy (DMT) | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Gender at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Gender at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Race at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Race at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients per United States Region at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients per United States Region at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Time since MS Diagnosis at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Time since MS Diagnosis at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients with Relapsing-remitting Multiple Sclerosis (MS) at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients with Relapsing-remitting MS at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients with Secondary Progressive MS at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients with Secondary Progressive MS at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients with Primary Progressive MS at Index Date by Vaccination Status | Index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients with Primary Progressive MS at Index Date by Prior DMT | Index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Mean Number of Comorbidities Within 12 Months Preceding Index Date by Vaccination Status | Within 12 months preceding index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Mean Number of Comorbidities Within 12 Months Preceding Index Date by Prior DMT | Within 12 months preceding index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients by Most Common Comorbidities (greater than 15%) Within 12 Months Preceding Index Date by Vaccination Status | Within 12 months preceding index date
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
  Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients by Most Common Comorbidities (greater than 15%) Within 12 Months Preceding Index Date by Prior DMT | Within 12 months preceding index date
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P. Index date was defined as the date of completion of full COVID-19 vaccination or the date of booster vaccination.
Number of Patients Treated with DMTs any Time Prior to Ofatumumab Initiation by Vaccination Status | Within 3 years of index date (defined as date of completion of full COVID-19 vaccination or date of booster vaccination)
  Three vaccination status levels were defined. Patients who were receiving ofatumumab at the time of:
  1. full COVID-19 vaccination and who received a booster vaccination (while continuing to receive ofatumumab), or
  2. booster vaccination but were not receiving ofatumumab at the time of full COVID-19 vaccination, or
  3. full COVID-19 vaccination but did not receive a booster vaccination or had discontinued ofatumumab before receipt of a booster vaccination.
  Full COVID-19 vaccination was defined as two doses of messenger ribonucleic acid (mRNA) vaccines (i.e., Pfizer, Moderna) or one dose of a single-dose adenoviral vaccine (i.e., Johnson and Johnson).
Number of Patients Treated with DMTs any Time Prior to Ofatumumab Initiation Categorized by Prior DMT | Within 3 years of index date (defined as date of completion of full COVID-19 vaccination or date of booster vaccination)
  DMTs included: DMT naïve, prior anti-CD20/sphingosine 1-phosphate (S1P) and prior non-anti-CD20/S1P.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States